CLINICAL TRIAL: NCT03514394
Title: DDBT Adapted Problem Solving Treatment for Primary Care
Acronym: PST-NA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Pat Arean, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00004236; 1P50MH115837-01 (NIH)
Record Dates: First submitted 2018-03-27; First posted 2018-05-02 (Actual); Results first posted 2022-08-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-07

CONDITIONS: Depression; PTSD
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Phase 1 will consist of observation and qualitative interviews; Phase two will consist of iterative design methods; phase three is a pilot randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Research Assistants and expert reviewers of therapy sessions will not be made aware of which condition the therapist is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual care administered for depression at clinic.
  Interventions: Behavioral: Usual Care
- Modified Behavioral Activation (Task Sharing) (Experimental): This intervention will be a modification of Behavioral Activation (BA), which is a behavioral intervention that identifies work, social, health, or family activities that patients have stopped engaging in because of their mood. Specifically, we will introduce a Task Sharing modification, which will allow clinicians and care managers to more efficiently share the tasks involved in BA. These modifications will be based on clinician and care manager feedback from Phases 1 and 2 of this study.
  Interventions: Behavioral: Modified Behavioral Activation (Task Sharing)

INTERVENTIONS:
Behavioral: Usual Care — The clinic's usual care includes counseling, substance use disorder treatment, peer support services, and some elements of traditional BA (not the modified BA).
  Arms: Usual Care
Behavioral: Modified Behavioral Activation (Task Sharing) — This intervention will include all core elements of Behavioral Activation (BA), which is a behavioral intervention that identifies work, social, health, or family activities that patients have stopped engaging in because of their mood. The intervention will also include a Task Sharing modification, which will allow clinicians and care managers to more efficiently share the tasks involved in BA.
  Arms: Modified Behavioral Activation (Task Sharing)

SUMMARY:
Evidence-based psychosocial interventions are rarely used in part because of their design complexity. Although many implementation frameworks do address the importance of EBPI characteristics, adapting and modifying EBPIs to enhance usability has not been a focus. User-centered design (UCD) approaches, which have been successful in creating hardware and software tools that are accessible and compelling to use, have the potential to modify EBPIs so that they are accessible and compelling to clinicians. We hypothesize that UCD driven modifications to EBPI usability (target mechanism) will result in enhanced clinician ability to deliver EBPI elements competently, and that better competence results in better patient reported outcomes. We will modify Behavioral Activation (BA), an EBPI often used in primary care, to function as a Task Sharing model between clinicians and care managers. Our specific aims are to (1) identify usability problems clinicians and care managers encounter with BA (2) create a clinician- and care manager-driven modification of BA and (3) compare the modified Task Sharing version of BA to usual care on usability, clinician competence, and patient reported outcomes.

DETAILED DESCRIPTION:
High quality delivery of evidence-based psychosocial interventions (EBPIs) in primary care medicine is a function of many variables, including clinician training and ready access to EBPI decision support. Importantly, quality is also driven by the clinician's ability to implement the therapeutic elements of EBPIs to fidelity and with competence. Even when clinicians undergo rigorous training, and find the intervention components useful in care, clinicians significantly drift from the original protocol because the processes, structure and elements of care frequently clash with clinician productivity and the shifting needs of the patient populations they serve. Clinicians in low resource settings like federally qualified health centers (FQHCs) report that while elements of EBPIs are important, their design is cumbersome, complex, overwhelming, inflexible, and minimize the nonspecific factors clinicians feel are crucial for quality delivery of care. In short, EBPIs demonstrate low usability (i.e., the extent to which a product can be used by specified users to achieve specified goals with effectiveness, efficiency, and satisfaction in a specified context of use. Although many implementation science (IS) frameworks do address the importance of EBPI characteristics, adapting and modifying EBPIs to enhance usability has not been a focus. User centered design (UCD) approaches, which have been successful in creating hardware and software tools that are accessible and compelling to use, have the potential to modify EBPIs so that they are accessible and compelling to clinicians. We hypothesize that UCD-driven modifications to EBPI usability will result in enhanced clinician ability to deliver EBPI elements competently (target), and that better competence results in better patient-reported outcomes. We will modify Behavioral Activation (BA) because it is the EBPI often used in primary care settings. To prepare for a larger trial to test hypotheses regarding the impact of EBPI usability on uptake, fidelity and competence, the aims of Project 002 R34 are:

Aim 1: Discover Phase (3 months). Using iterative and participatory methods, we will interview up to 15 clinicians from FHQCs affiliated with the WWAMI region Practice Research Network (WPRN, a collaborative group of primary care practices through the states of Washington, Wyoming, Alaska, Montana and Idaho to facilitate innovative community-based research), and observe them in routine practice to identify usability challenges. Contribution to the Center: Data from this phase will be used to inform the Typology of EBPI Targets.

Aim 2: Design/Build Phase (6 months) After identification of potential targets, the research team will work via Zoom teleconferencing with the original clinicians from the discover phase and 0-5 new clinicians to engage in a rapid cycle of iterative prototype development and testing (e.g., storyboarding, paper prototypes) of BA modifications. The build of these modifications will include the development of intervention prototypes for user testing and refinement with input from these care managers. Contribution to the Center: Data from this phase will be used to inform the Matrix of EBPI Modifications.

Aim 3: Test Phase (15 months). We will test and compare the BA modification (Task Sharing) to usual care in a small non-randomized trial. We will assign all provider teams (therapist & care manager(s)) in the clinic to use Task Sharing with their patients. We will then compare patient outcomes for those receiving Task Sharing vs. patients receiving usual clinic care. H1: Modifications developed in the Design/Build phase for targets identified in the Discover Phase will result in better usability (System Usability and User Burden Scales) compared to usual care. H2: Task Sharing will be more effective than usual care on improving clinical outcomes of functional disability (Sheehan Disability Scale [SDS]), change in depression symptoms over time (PHQ-9 total score), and change in anxiety symptoms over time (GAD-7 total score).

ELIGIBILITY:
Inclusion Criteria:

* Primary care patient in rural MT and WY; Speaks English; Patient Health Questionnaire - 9 > 10.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, PhD, Principal Investigator — UWMC Psychiatry
Locations (1):
- Big Horn Valley Health Center, Hardin, Montana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the UW ALACRITY Center once it is collected and analyzed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available January 2022
Access Criteria: All interested parties may contact Dr. Renn for access to data. Dr. Renn will review all requests and facilitate data use agreements and data access.

REFERENCES:
- [Derived] Lyon AR, Munson SA, Renn BN, Atkins DC, Pullmann MD, Friedman E, Arean PA. Use of Human-Centered Design to Improve Implementation of Evidence-Based Psychotherapies in Low-Resource Communities: Protocol for Studies Applying a Framework to Assess Usability . JMIR Res Protoc. 2019 Oct 9;8(10):e14990. doi: 10.2196/14990. PMID 31599736

RESULTS

PARTICIPANT FLOW:
Groups:
- Task Sharing - Patients; Task Sharing - Clinicians: Task sharing is a modified version of a depression treatment called Behavioral Activation, which allows therapists and care managers to more efficiently share the tasks involved in patient care.
Period: Overall Study
Arm/Group | Usual Care | Task Sharing - Patients | Task Sharing - Clinicians
Started | 17 | 16 | 11
Completed | 17 | 16 | 10
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants in the Usual Care arm include 17 patients. Participants in the Task Sharing Arm include 16 patients and 11 clinicians. The task sharing arm is broken up into two columns to separate clinician and patient participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Task Sharing - Patients | Task Sharing - Clinicians | Total
Number analyzed (Participants) | 17 | 16 | 11 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One clinician in the Task Sharing arm did not contribute age data.
  years
    number analyzed (Participants) | 17 | 16 | 10 | 43
    (all) | 37.9 (15.0) | 39.5 (13.9) | 39.3 (9.6) | 38.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One clinician participant in the task sharing arm did not contribute demographic data.
  Participants
    number analyzed (Participants) | 17 | 16 | 10 | 43
    Female | 14 | 14 | 9 | 37
    Male | 3 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 16 | 10 | 40
  Unknown or Not Reported | 3 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 6 | 2 | 12
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 10 | 8 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — Population: Clinicians were not administered the PHQ, so they are left blank here. Only 13 of the participants in the intervention condition responded to enough items on the PHQ at baseline to compute their score.
  units on a scale
    number analyzed (Participants) | 17 | 13 | 0 | 30
    (all) | 18.4 (7.5) | 11.0 (6.9) |  | 15.2 (8.0)
Generalized Anxiety Disorder (7-item) Scale (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — Population: Clinicians did not respond to this measure, so they are not included here. Only 13 participants in the intervention condition responded to this measure.
  units on a scale
    number analyzed (Participants) | 17 | 13 | 0 | 30
    (all) | 14.6 (6.2) | 8.1 (6.7) |  | 11.8 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: 9 item patient self report measure of mood, where each item as rated on a 0 (no problem) to 3 (every day) scale. Total scores range from 0 - 27. Higher scores indicate increased depression, a score of 10 or greater is considered to be clinical depression. Data points were collected from each individual multiple times across the course of the study. For comparisons we conducted a multiple case study design examining each person's individual trajectory. The means and standard deviations reported are for all available observations stratified by condition.
Time Frame: Patient participants will complete the PHQ-9 at baseline and weekly for 10 weeks, single value calculated averaging across all available observations.
Population: Sample sizes were too small to appropriately run any tests of statistical significance. Data points were collected from each individual multiple times across the course of the study. For comparisons we conducted a multiple case study design examining each person's individual trajectory. The means and standard deviations above are for all available observations stratified by condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Task Sharing - Patient: Task sharing is a modified version of a depression treatment called Behavioral Activation, which allows therapists and care managers to more efficiently share the tasks involved in patient care.
Arm/Group | Usual Care | Task Sharing - Patient
Number analyzed (Participants) | 17 | 16
score on a scale | 13.3 (6.6) | 10.7 (6.8)

2. Primary Outcome: Generalized Anxiety Disorder (7-item) Scale (GAD-7)
Description: A 7-item screener for generalized anxiety. It consists of items related to GAD. Participants rate on a scale of 0-3 how much they have experienced in the last two weeks. Total scores range from 0 - 21. The scale is a valid screener for GAD. High scores indicate higher anxiety symptom severity. Data points were collected from each individual multiple times across the course of the study. For comparisons we conducted a multiple case study design examining each person's individual trajectory. The means and standard deviations reported are for all available observations stratified by condition.
Time Frame: Patient participants will complete the GAD-7 at baseline and weekly for 10 weeks, single value calculated averaging across all available observations.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Task Sharing - Patient
Number analyzed (Participants) | 17 | 16
score on a scale | 10.2 (6.7) | 8.1 (5.3)

3. Secondary Outcome: Acceptability Intervention Measure (AIM)
Description: This is a four item measure of intervention acceptability, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. Total scores are calculated taking the mean of the four items, reporting a range of 1 - 5.
Time Frame: Clinician participants will complete the AIM at baseline and 3-month follow-up.
Population: Clinicians in the task sharing arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Task Sharing: Task sharing is a modified version of a depression treatment called Behavioral Activation, which allows therapists and care managers to more efficiently share the tasks involved in patient care.
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 10
score on a scale
  Baseline: number analyzed (Participants) | 0 | 8
  Baseline |  | 4.6 (0.5)
  3-month Follow Up |  | 4.5 (0.5)

4. Secondary Outcome: User Burden Scale
Description: The User Burden Scale is a 26-item scale that assesses six domains of user burden: use, physical burden, time/social burdens, mental/emotional burden, privacy concerns and financial burdens. The scale is calculated item measure of perceived burden of use that covers 6 domains: difficulty of use, emotional burden, physical burden, time and social burden, financial burden and privacy. Each item is rated on a 04- scale, with a maximum score of 104 (high burden) and minimum score of 0 (low burden). We will compare the ratings of intervention burden between groups to determine if the new intervention is considered less burdensome than the traditional model.
Time Frame: Clinician participants will complete the UBS at baseline and 3-month follow-up.
Population: Clinicians in the task sharing arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 10
score on a scale
  Baseline: number analyzed (Participants) | 0 | 8
  Baseline |  | 5.0 (5.2)
  3-month Follow Up |  | 5.0 (6.0)

5. Secondary Outcome: Time to Certification
Description: We will record the number of hours needed for clinicians in each group to be trained in their assigned intervention.
Time Frame: Hours toward certification will be collected over a three month period.
Population: No data displayed because outcome measure data was not collected therefore zero total participants analyzed.
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Skill Drift Using the PST Adherence Checklist
Description: This is a 20 item scale, where each item rates clinician competencies in the delivery of PST, using a 0 (not competent) to 5 (expert level) scale. Higher scores indicate greater competence. IN this use case, we will be measuring the time to which clinicians receive their first score below 3 (average) on the PST Adherence Checklist
Time Frame: We will rate nine therapy sessions per clinician over a six month period.
Population: No data displayed because outcome measure data was not collected therefore zero total participants analyzed.
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: System Usability Scale
Description: This is a 10-item scale with each item ranked on a five point system of low to high usability. The scale score is calculated by adding the item scores and multiplying by 2.5. This is your total score and can range from 0 - 100. A score of 68 or better is considered to be above average usability. A score less than 68 is considered to be poor usability. In this study, a score of 80 or more is considered our cut off for high usability.
Time Frame: Clinician participants will complete the SUS at baseline and 3-month follow-up
Population: Clinicians in the task sharing arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 10
score on a scale
  Baseline: number analyzed (Participants) | 0 | 8
  Baseline |  | 73.4 (9.3)
  3-month Follow-Up |  | 73.0 (8.5)

8. Secondary Outcome: Intervention Appropriateness Measure (IAM)
Description: This is a four item measure of intervention appropriateness, where each item is rated on a 1-5, with 1 = not at all acceptable and 5 = very acceptable. High scores (min: 1, max:5) indicate higher levels of appropriateness. Total scores are calculated taking the mean of the four items, reporting a range of 1 - 5.
Time Frame: Clinician participants will complete the IAM at baseline and 3-month follow-up
Population: Clinicians in the task sharing arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 9
score on a scale
  Baseline: number analyzed (Participants) | 0 | 8
  Baseline |  | 4.7 (0.5)
  3-month Follow-Up |  | 4.3 (0.5)

9. Secondary Outcome: Feasibility of Intervention Measure (FIM)
Description: This is a four-item measure of intervention feasibility, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. Higher scores indicate higher levels of feasibility. Total scores are calculated taking the mean of the four items, reporting a range of 1 - 5.
Time Frame: Clinician participants will complete the FIM at baseline and 3-month follow-up
Population: Clinicians in the task sharing arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Task Sharing
Number analyzed (Participants) | 0 | 10
score on a scale
  Baseline: number analyzed (Participants) | 0 | 8
  Baseline |  | 4.6 (0.4)
  3-month Follow-Up |  | 4.4 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entirety of time patients were in the study from baseline to 10 week follow-up.
Groups:
- Usual Care - Patients: Usual care administered for depression at clinic.
Arm/Group | Usual Care - Patients | Task Sharing - Patients
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT03514394/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT03514394/ICF_001.pdf